CLINICAL TRIAL: NCT00190099
Title: Dexamethasone-Eluting Stent in Acute Coronary Syndrome to Prevent Restenosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FEMH-93005
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2005-11-18 (Estimated); Status verified 2004-12

CONDITIONS: Vessel Restenosis
Keywords: In-stent restenosis,; Drug eluting stent,; dexamethasone,; Acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

INTERVENTIONS:
Device: Dexamethasone-Eluting Stent

SUMMARY:
The major obstacle of the long- termed success of percutaneous coronary intervention (PCI) is the restenosis. Restenosis results from complex pathophysiological response of the vascular tissue to the balloon injury. In the pre-stent era, 80% of it was attributed to vascular recoil. However, by way of the mechanical support of metallic stent, recoil is no more the major reason of restenosis. About 80 % of In-stent restenosis resulted from intimal hyperplasia.

The mechanism of the Intra-stent restenosis included 4 stages. First stage comprised the first 3 days after balloon injury, when the inflammatory reaction is most severe throughout the course. At that time, anti-inflammatory drug as steroid wuold be helpful to prevent the course of restenosis. Until the end of the third week, smooth muscle cells migrate and then proliferate in the second and the third stage, and the key effort to prevent restenosis right now is inhibition of cell cycle. Intravascular radiotherapy (so called Brachytherapy) and stent-based drug elution target upon them. Among them, rapamycin and paclitaxel proved to be effective both in animal and human experience. The last stage is re-epithelization, estrogen could promote the process and was considered to be effective in this stage.

Stent-based elution of corticosteroid, despite of its feasibility and safety, was not as effective as other anti-proliferation agent ( eg. Rapamycin etc). The major reason might be the patient group with coronary artery disease is a heterogenous one.

We believe if we applied corticosteroid over the patient with elevated inflammatory parameters, i.e. acute coronary syndrome (ACS) the effect of anti-restenosis would be obvious.

In this study, by a special-designed, phosphorylcholine-coated stent, dexamethasone could be readily absorbed and then gradually released locally even 4 weeks after deployment.

We expected a reduction of In-stent restenosis in ACS patient by the method with no or few systemic adverse effect of steroid; and angiographic follow-up as well as intra-vascular ultrasound assessment would be performed according to pur protocol.

DETAILED DESCRIPTION:
The major obstacle of the long- termed success of percutaneous coronary intervention (PCI) is the restenosis. Restenosis results from complex pathopysiological response of the vascular tissue to the balloon injury. In the pre-stent era, 80% of it was attributed to vascular recoil. However, by way of the mechanical support of metallic stent, recoil is no more the major reason of restenosis. About 80 % of In-stent restenosis resulted from intimal hyperplasia.

The mechanism of the Intra-stent restenosis included 4 stages. First stage comprised the first 3 days after balloon injury, when the inflammatory reaction is most severe throughout the course. At that time, anti-inflammatory drug as steroid would be helpful to prevent the course of restenosis. Until the end of the third week, smooth muscle cells migrate and then proliferate in the second and the third stage, and the key effort to prevent restenosis right now is inhibition of cell cycle. Intravascular radiotherapy (so called Brachytherapy) and stent-based drug elution target upon them. Among them, rapamycin and paclitaxel proved to be effective both in animal and human experience. The last stage is re-epithelization, estrogen could promote the process and was considered to be effective in this stage.

Stent-based elution of corticosteroid, despite of its feasibility and safety, was not as effective as other anti-proliferation agent ( eg. Rapamycin etc). The major reason might be the patient group with coronary artery disease is a heterogenous one.

We believe if we applied corticosteroid over the patient with elevated inflammatory parameters, i.e. acute coronary syndrome (ACS) the effect of anti-restenosis would be obvious.

In this study, by a special-designed, phosphorylcholine-coated stent, dexamethasone could be readily absorbed and then gradually released locally even 4 weeks after deployment.

We expected a reduction of In-stent restenosis in ACS patient by the method with no or few systemic adverse effect of steroid; and angiographic follow-up as well as intra-vascular ultrasound assessment would be performed according to pur protocol.

ELIGIBILITY:
Inclusion Criteria:

* ACS patient

Exclusion Criteria:

-

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2003-01; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: A H Li, MD, Principal Investigator — Far Eastern Memorial Hospital